CLINICAL TRIAL: NCT00323102
Title: Phase IV, Double-Blind, Multi-Center, Randomized, Cross-Over Study to Compare 0.10 Mmol/kg of MultiHance With 0.10 Omniscan in Magnetic Resonance Imaging (MRI) of the Brain
Brief Title: A Study Comparing Two Magnetic Resonance Imaging (MRI) Contrast Agents in MRI of the Brain
Acronym: ENHANCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: MH 130
Record Dates: First submitted 2006-05-05; First posted 2006-05-09 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2008-01

CONDITIONS: Brain Pathology
MeSH Terms: interventions — gadobenic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Multihance

SUMMARY:
This study aims at a direct comparison between Multihance and a validated comparator like Omniscan in a cross-over individual design in patients with brain tumors to confirm the superior overall diagnostic performance of MuliHance for this indication

ELIGIBILITY:
Inclusion Criteria:

* 18 yrs of age or older; provide written informed consent; scheduled to undergo MRI; willing to undergo 2 MRI exams within 14 days

Exclusion Criteria:

* Known allergy to one or more ingredients in the test agents; severe CHF (Class IV); suffered stroke one year ago; pregnancy or lactating females; contraindications to MRI; severe claustrophobia; scheduled to receive surgery prior to or between the two MRI exams, or steroids or radiosurgery between the two MRI exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114
Dates: Start 2006-05; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Superiority of Multihance in terms of by-patient global diagnostic performance | immediately post dose

SECONDARY OUTCOMES:
To compare the two products in terms of by patients global performance for border delineation of lesions; contrast of lesions | immediately post dose
To compare the two products in terms of global changes in lesion count; To compare the two products in terms of changes from pre to post dose in signal intensity | immediately post dose

CONTACTS AND LOCATIONS:
Overall Officials: Barry Hogstrom, M. D., Study Director — Bracco Diagnostics, Inc
Locations (1):
- Bracco Diagnostics, Inc., Princeton, New Jersey, United States